CLINICAL TRIAL: NCT02493439
Title: A Positive Activity Intervention to Promote Optimism and Psychological Wellbeing in Romanian Immigrants
Brief Title: A Positive Activity Intervention to Promote Wellbeing in Romanian Immigrants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJaumeI013
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Immigrants
Keywords: Best Possible Self; Positive Psychology; Romanian Immigrants; Optimism; Future Thinking
MeSH Terms: interventions — Activities of Daily Living

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best Possible Self (Experimental): Participants are asked to write and imagine about a future in which they have reached all their goals in four different domains: personal, professional, social and health. The participants are instructed to practice the BPS intervention for a month, 5 minutes/day.
  Interventions: Behavioral: Best Possible Self
- Daily Activities (Placebo Comparator): Participants are asked to think and write about the activities carried out in the last 24 hours. The participants are instructed to practice the Daily Activities exercise for a month, 5 minutes/day.
  Interventions: Behavioral: Daily Activities

INTERVENTIONS:
Behavioral: Best Possible Self
  Arms: Best Possible Self
Behavioral: Daily Activities
  Arms: Daily Activities

SUMMARY:
This study aims to test the efficacy of an intervention focused on promoting positive emotions (Best Possible Self - BPS) to improve the psychological wellbeing of Romanian immigrants living in Spain. It is hypothesized that the BPS intervention will significantly improve a series of positive mental health outcomes, i.e., optimism, future expectancies, and affect, compared to the Control group.

DETAILED DESCRIPTION:
Previous studies have shown that groups of immigrants may face a series of problems unique to the process of immigration, such as working, legal, social, and mental and physical health problems.

BPS is a guided imagery exercise that requires participants to envision themselves in the future, achieving desired goals in different areas of their lives. This exercise has shown efficacy improving optimism, future expectancies and positive affect compared to a control condition, in general population. Taking into account the prior literature, the aim of the present study is to carry out a randomized controlled study in order to replicate the findings about the effects of BPS on optimism, mood and affect in an immigrant population. The design employed in this study is similar to the used in other studies.

ELIGIBILITY:
Inclusion Criteria:

* Romanian immigrant in Spain
* Sign a consent form stating their willingness to participate

Exclusion Criteria:

* Presence of severe physical illness
* Presence of severe psychological disorder
* Be currently involved in another psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Subjective Probability Task | 1 month
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 and 0.91, respectively)

SECONDARY OUTCOMES:
Positive and Negative Affect Scale | 1 month
  This measure analyzes the levels of positive (PA) and negative affect (NA). The instrument consists of 20 items, 10 for each level of affect. Participants rate on a 5-point scale (Not at all - Extremely).
Beck Depression Inventory II | 1 month
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and test-retest reliability of around 0.8.
Overall Anxiety Severity and Impairment Scale | 1 month
  OASIS is a brief instrument consisting of 5 items that measure the frequency and severity of anxiety, as well as the level of avoidance and work/school/home and social interference that anxiety produces.
Dysfunctional Attitudes Scale | 1 month
Difficulties in Emotion Regulation Scale | 1 month
Life Orientation Test | 1 month
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 and 0.91, respectively).
Hope Scale | 1 month
Quality of Life Index | 1 month
  It consists of 10 items that evaluate perceived well-being in different areas (physical, psychological/emotional, occupational functioning, interpersonal functioning, among others)
Ryff Scales of Psychological Well-Being | 1 month

OTHER OUTCOMES:
Self Concordance Motivation | baseline
  This questionnaire assess extrinsic and intrinsic motivation to practice the imagery exercise, rated on a 9-point scale ranging from 1 "not at all for this reason" to 9 "completely for this reason". SCM has been correlated withparticipants' frequency of practicing a daily imagery exercise and with self-reported imagery performance, a key aspect in self-applied interventions.
Multidimensional Scale of Perceived Discrimination | baseline
  This scale is made up of 20 items that measure four aspects of perceived discrimination: blatant group discrimination, subtle group discrimination, blatant individual discrimination and subtle individual discrimination.
Social Support | baseline
  This scale is an adapted version of the questionnaire designed by Gonzalez-Castro and Ubillos (2011). This questionnaire measures the social support received from other Romanians in Spain and from the Spanish people, in three areas: tangible social support (support in leisure activities), emotional support (care, love) and informational and instrumental support (help in addressing problems). In addition, the questionnaire measures the support received from those who live in the country of origin of the immigrant (1 = never receives support, 4 = receives a lot of support).

CONTACTS AND LOCATIONS:
Overall Officials: Azucena García-Palacios, PhD, Principal Investigator — Universitat Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

REFERENCES:
- [Background] Meevissen YM, Peters ML, Alberts HJ. Become more optimistic by imagining a best possible self: effects of a two week intervention. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):371-8. doi: 10.1016/j.jbtep.2011.02.012. Epub 2011 Mar 2. PMID 21450262
- [Background] Peters ML, Flink IK, Boersma K, Linton SJ. Manipulating optimism: can imagining a best possible self be used to increase positive future expectancies? Journal of Positive Psychology 5: 204-211, 2010.
- [Background] MacLeod, Byrne, & Valentine (1996). Affect, emotional disorder, and future-directed thinking. Cognition & Emotion 10: 69-86.
- [Background] Molero, F., Recio, P., García-Ael, C., Fuster, M. J., & Sanjuán, P. (2013). Measuring dimensions of perceived discrimination in five stigmatized groups. Social indicators research, 114(3), 901-914.
- [Background] Gonzalez-Castro JL, Ubillos S. Determinants of psychological distress among migrants from Ecuador and Romania in a Spanish city. Int J Soc Psychiatry. 2011 Jan;57(1):30-44. doi: 10.1177/0020764009347336. PMID 21252354
- [Background] Renner F, Schwarz P, Peters ML, Huibers MJ. Effects of a best-possible-self mental imagery exercise on mood and dysfunctional attitudes. Psychiatry Res. 2014 Jan 30;215(1):105-10. doi: 10.1016/j.psychres.2013.10.033. Epub 2013 Nov 1. PMID 24252218
- [Background] Sheldon, K. M., & Lyubomirsky, S. (2006). How to increase and sustain positive emotion: The effects of expressing gratitude and visualizing best possible selves. The Journal of Positive Psychology, 1(2), 73-82.